CLINICAL TRIAL: NCT03534544
Title: Patient and Parent Preferences for an On-Body Automated Insulin Delivery System
Status: Completed | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lori Laffel, Chief, Pediatric, Adolescent, and Young Adult Section; Co-Head, Section on Clinical, Behavioral and Outcomes Research, Joslin Diabetes Center
Other Study IDs: CHS2018-05; DP3DK113511 (NIH)
Record Dates: First submitted 2018-04-20; First posted 2018-05-23 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: artificial pancreas; pediatric; parents; adherence
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to learn more about patient and family preferences regarding use of advanced diabetes technologies. Young persons with type 1 diabetes (ages 8-25) and parents of young persons with type 1 diabetes will complete one study visit involving a semi-structured interview and surveys. The results of the study will be used to assist in the design of a new automated insulin delivery system.

DETAILED DESCRIPTION:
Type 1 diabetes remains the most common chronic disease of childhood and affects millions of children and adults globally. The minority of persons with type 1 diabetes achieve the recommended glycemic targets. Currently approved and unapproved automated insulin delivery systems require patients to carry and wear multiple devices (pumps, tubing, blood glucose meters, mobile devices, etc.). There is a need to design automated insulin delivery systems that reduce the burden of diabetes management for young persons and their families in an effort to improve glycemic control as well as other biomedical and psychosocial outcomes.

The purpose of this study is to conduct separate semi-structured interviews with young persons with type 1 diabetes and parents of youth with type 1 diabetes (not necessarily the parents of the youth participants) regarding their preferences for an automated, on-body insulin delivery system. Youth and parents will also complete short surveys related to perceived burden of diabetes self-care, quality of life, acceptance of diabetes, and worries about hypoglycemia. The feedback received from the interviews and surveys will help inform the design of a new on-body automated insulin delivery system.

ELIGIBILITY:
Inclusion Criteria:

* Young persons (ages 8-25 years) with type 1 diabetes for 1 year or longer
* Parents of young persons with type 1 diabetes

Exclusion Criteria:

* None

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be recruited from the clinic populations of the 2 study sites.
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Youth and parent preferences for automated insulin delivery systems | 1 day
  Semi-structured interviews with young persons with type 1 diabetes and parents; interviews will be transcribed and analyzed to derive central themes; this is a qualitative outcome

SECONDARY OUTCOMES:
Diabetes burden | 1 day
  Problem Areas in Diabetes survey - Pediatric version (PAID-Peds) and Parent revised version (PAID-PR)
  * PAID-Peds: 20 items, PAID-PR: 18 items
  * Possible score: 0-100
  * Higher score indicates more burden
Worries about hypoglycemia | 1 day
  Fear of Hypoglycemia survey - Worry Scale
  * 15 items
  * Possible score: 0-100
  * Higher score indicates more worry about hypoglycemia
Diabetes acceptance | 1 day
  Accepting Diabetes and Personal Treatment (ADAPT) survey
  * 24 items
  * Scoring methodology will be established with data from this study
Quality of life | 1 day
  5-Item World Health Organization (WHO-5) Well-Being Index
  * 5 items
  * Possible score: 0-100 (percentage score)
  * Higher score indicates better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Lori Laffel, MD, MPH, Principal Investigator — Joslin Diabetes Center; Stuart Weinzimer, MD, Principal Investigator — Yale University; Eyal Dassau, PhD, Principal Investigator — Harvard University
Locations (2):
- United States (2):
  - Yale University School of Medicine, New Haven, Connecticut
  - Joslin Diabetes Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided
Qualitative data may be available after removal of all personal identifiers.

REFERENCES:
- [Result] Commissariat PV, Volkening LK, Butler DA, Dassau E, Weinzimer SA, Laffel LM. Innovative features and functionalities of an artificial pancreas system: What do youth and parents want? Diabet Med. 2021 Oct;38(10):e14492. doi: 10.1111/dme.14492. Epub 2021 Jan 20. PMID 33290599
- [Result] Commissariat PV, Roethke LC, Finnegan JL, Guo Z, Volkening LK, Butler DA, Dassau E, Weinzimer SA, Laffel LM. Youth and parent preferences for an ideal AP system: It is all about reducing burden. Pediatr Diabetes. 2021 Nov;22(7):1063-1070. doi: 10.1111/pedi.13252. Epub 2021 Aug 9. PMID 34324772